CLINICAL TRIAL: NCT07104526
Title: Evaluation of the Efficacy and Safety of Low-Dose Propranolol Combined With Intralesional Bleomycin for Infantile Hemangioma: A Randomized Controlled Trial
Brief Title: Low-Dose Propranolol and Bleomycin for Infantile Hemangioma (IH)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wuhan Integrated Traditional Chinese and Western Medicine Hospital (Other)
Responsible Party: Principal Investigator, Bin Zhou, Principal investigator, Wuhan Integrated Traditional Chinese and Western Medicine Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023R064-E01
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Infantile Hemangioma (IH)
MeSH Terms: conditions — Hemangioma, Capillary | interventions — Propranolol; Bleomycin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Combination Therapy Group (Experimental): Participants received oral propranolol hydrochloride solution at a dose of 1 mg/kg/day (in two divided doses) for 6 months, combined with intralesional injections of bleomycin. Bleomycin injections were administered once a month for up to 6 months.
  Interventions: Drug: Propranolol + Bleomycin
- Active Comparator: Propranolol Monotherapy Group (Active Comparator): Participants received oral propranolol hydrochloride solution at a dose of 1 mg/kg/day (in two divided doses). The total treatment duration was 6 months.
  Interventions: Drug: Propranolol

INTERVENTIONS:
Drug: Propranolol + Bleomycin — Oral propranolol at 1 mg/kg/day for 6 months plus intralesional bleomycin (1 mg/mL solution) injected once monthly. The bleomycin dose was 0.2-0.5 mg per injection site, not exceeding a total of 1 mg/kg per session or a cumulative dose of 10 mg.
  Arms: Experimental: Combination Therapy Group
Drug: Propranolol — Oral propranolol hydrochloride solution administered at a dose of 1 mg/kg/day for 6 months.
  Arms: Active Comparator: Propranolol Monotherapy Group

SUMMARY:
This is a prospective, randomized controlled trial designed to evaluate the efficacy and safety of low-dose oral propranolol (1 mg/kg/day) combined with monthly intralesional bleomycin injections versus low-dose propranolol monotherapy for the treatment of infantile hemangioma (IH). A total of 260 infants were randomized to either the combination group or the control group. The study aims to determine if the combination therapy offers superior clinical outcomes, including faster regression, better color resolution, and reduced scarring over a 6-month treatment period.

DETAILED DESCRIPTION:
Infantile hemangioma (IH) is the most common benign vascular tumor in infancy. While oral propranolol is the first-line systemic therapy, its efficacy can be limited or slow for certain IHs. Intralesional bleomycin offers a targeted local therapy. This study investigates whether combining low-dose propranolol with local bleomycin injections can enhance therapeutic effects while maintaining a good safety profile. This prospective, randomized, controlled, open-label trial with blinded outcome assessment enrolled 260 infants with IH. Participants were randomly assigned to receive either oral propranolol (1 mg/kg/day) plus monthly intralesional bleomycin (Combination Group) or oral propranolol (1 mg/kg/day) alone (Control Group) for 6 months. The primary objective is to compare the clinical therapeutic effect between the two groups at 6 months. Secondary objectives include evaluating early tumor response, changes in tumor volume and color, long-term scar formation, and the incidence of adverse events. The findings aim to provide robust evidence for a potentially more effective combination treatment strategy for IH.

ELIGIBILITY:
Inclusion Criteria:

* Age ≤12 months.
* Clinically and/or imaging-diagnosed infantile hemangioma requiring treatment.
* No prior treatment for IH.
* Guardians willing to comply with the study protocol and provide informed consent.

Exclusion Criteria:

* Known hypersensitivity to propranolol or bleomycin.
* Congenital or mixed hemangiomas distinct from IH.
* Significant cardiopulmonary, hepatic, or renal dysfunction.
* Presence of other severe systemic diseases.
* PHACE syndrome or major congenital anomalies that could interfere with treatment or assessment.

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 260 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Clinical Therapeutic Effect | 6 Months
  Categorized as Complete Regression (>95% volume reduction), Marked Effectiveness (≥75% to 95% volume reduction), Effective (30% to <75% reduction), or Ineffective (<30% reduction). The primary measure is the rate of participants achieving Complete Regression or Marked Effectiveness.

SECONDARY OUTCOMES:
Early Tumor Surface Atrophy | 24 hours after the first treatment
  Assessed by comparing photographs and graded as Obvious Atrophy, Mild Atrophy, or No Obvious Change.
Change in Hemangioma Color Score | Baseline, 6 Months
  Rated on a 4-point subjective scale (0-3) based on standardized digital photographs, where a lower score indicates color closer to normal skin. The change from baseline is assessed.
Change in Tumor Volume | Baseline, 6 Months
  Measured in cubic centimeters (cm³) using high-frequency color Doppler ultrasound (Volume = length × width × height × 0.52). The change from baseline is assessed.
Vancouver Scar Scale (VSS) Score | 6 Months
  Assessed at the former hemangioma site. The VSS evaluates pigmentation, vascularity, pliability, and height, with a total score from 0 (normal skin) to 13 (worst scar). Lower scores indicate better outcomes.
Incidence of Adverse Events | Through study completion (6 months)
  Number and type of local and systemic adverse events reported by guardians or observed clinically (e.g., injection site reactions, bradycardia, hypoglycemia, sleep disturbances).

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan Children's Hospital, Wuhan, Hubei, China